CLINICAL TRIAL: NCT02474160
Title: Patient-Derived Models Tissue Procurement Protocol for the National Cancer Institute (NCI)
Brief Title: Collection and Storage of Tissue and Blood Samples From Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute LAO (Unknown)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: NCI-2015-00863; NCI-2015-00863 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P9846; P9846_R02PAPPHOLD01; 9846 (Other: National Cancer Institute LAO); 9846 (Other: CTEP); UM1CA186689 (NIH); UM1CA186691 (NIH); UM1CA186704 (NIH); UM1CA186709 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (tissue and blood procurement): Tumor tissue and blood samples are procured during procedures that are required for the patients' clinical management and stored via xenograft (transplant to another species) models or in vitro cell culture for future analysis.
  Interventions: Other: Cytology Specimen Collection Procedure

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Procurement of tissue and blood samples
  Other Names: Cytologic Sampling

SUMMARY:
This study collects and stores tissue and blood samples from patients with cancer. Collecting and storing samples of tissue and blood from patients with cancer to study in the laboratory may help scientists create new and better models to learn about cancer and to test new cancer drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To procure biologic tissues and materials to generate preclinical models of cancer.

OUTLINE: This is an observational study.

Tumor tissue and blood samples are procured during procedures that are required for the patients' clinical management and will be stored via xenograft (transplant to another species) models or in vitro cell culture for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 2 months of age who are being evaluated, treated, or enrolled in a clinical trial for cancer at participating sites
* Patients with a histologically or cytologically confirmed diagnosis of cancer
* Patients without histologically or cytologically confirmed diagnosis of cancer, but for whom approval has been requested and received from the coordinating site study coordinator

  * Requests for coordinating site approval should only be made if the patient's existing work-up at the time of the request demonstrates a combination of two or more of the following indicating the greater likelihood of a cancerous process in the assessment of the treating physician:

    * Radiographic imaging (computed tomography [CT], magnetic resonance imaging [MRI], etc.)
    * Elevated tumor markers
    * Clinical symptoms
    * Documented risk factors, known genetic changes (mutation, deletion, fusion, etc.), and/or known familial cancer history or syndrome
    * Complete blood count (CBC) w/differential indicative of a probable hematologic malignancy
  * If the patient will be undergoing surgical resection at a later time and will be accessible to approach for study participation at that time, resected material following cancer diagnosis confirmation is preferred
  * Important: Additional medical, genetic and/or demographic work-up should not be obtained solely for determination of eligibility for protocol 9846 by these criteria. Once available, final histology must be confirmed to the coordinating site detailing the cancer diagnosis for patients enrolled based on the above criteria
* Patients with a newly diagnosed primary and/or metastatic solid tumor or hematologic malignancy for which they have not yet received treatment
* Patients with a solid tumor or hematologic malignancy that is recurrent, newly metastasized, or progressing while on treatment indicated by:

  * Radiographic evidence of tumor growth, re-growth, and/or new metastases, OR
  * Documentation by the treating physician of clinical disease progression, OR
  * CBC w/differential and/or flow cytometry for hematologic malignancies
* Patients currently undergoing treatment (adjuvant, neoadjuvant, etc.)

  * Specimen collection should occur as distant in time from the most recent drug administration as possible (e.g., after completion of a treatment cycle and immediately prior to initiation of the next cycle)
  * Specimens should not be collected from patients between doses within a single treatment cycle
  * Confirmation of viable residual malignancy and/or < 90% tumor necrosis, fibrosis, or hemorrhage must be confirmed to the National Cancer Institute (NCI) coordinating site, as indicated in the final post-operative/post-procedure pathology and/or flow cytometry report
* Patients with ongoing partial response (PR) or stable disease (SD) are eligible

  * Confirmation of viable malignancy and/or < 90% tumor necrosis, fibrosis, or hemorrhage must be confirmed to the NCI coordinating site, as indicated in the final post-operative/post-procedure pathology and/or flow cytometry report
* Ability to understand and willingness to sign a written informed consent document indicating their willingness to have their tissue or biologic fluid specimens used for research as outlined in this protocol

  * For pediatric patients, ability and willingness to assent to participation, using an explanation that is understandable/age appropriate, as well as receiving parental permission. Signature requirements for pediatric patients can be adjusted based on local guidelines

Exclusion Criteria:

* Patients with cancer-like syndromes and/or blood disorders such as systemic mastocytosis, Langerhans cell histiocytosis, chronic eosinophilic leukemia/hypereosinophilic syndrome, lymphomatoid granulomatosis, or monoclonal gammopathy of undetermined significance (MGUS)
* Patients with invasive fungal infections
* Patients with active and/or uncontrolled bacterial, fungal, or viral infections or who are still recovering from an infection

  * Actively febrile patients with uncertain etiology of febrile episode
  * All antibiotics prescribed for the treatment of a bacterial infection should be completed at least 1 week (7 days) prior to collection

    * Patients with a hematologic malignancy who are treated with an antibiotic, anti-fungal, and/or anti-viral medication for an active infection who then remain on the treatment for prophylaxis following resolution of the infection as assessed by the treating physician are not excluded
  * No recurrence of fever or other symptoms related to infection for at least 1 week (7 days) following completion of antibiotics
  * Patients receiving antibiotics, antifungals, and/or antivirals for prophylaxis are permissible
  * Antibiotics being administered topically at a location distant from the planned tissue collection site or eye drops for a localized infection are permissible
* Patients with human immunodeficiency virus (HIV), active or chronic hepatitis (i.e., quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA]) or known history of HCV, HBV, or HIV; testing for HBV, HCV, HIV or other infections for eligibility will be performed only if clinically indicated
* Patients with hepatitis A as indicated by anti-hepatitis A virus (HAV) IgM reactivity

  * Patients that are anti-HAV IgG reactive only are eligible
* Specimen collections from patients with benign tumors including but not limited to desmoid tumors, carcinoma in situ, or ongoing evidence of complete disease response (CR)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing evaluation and/or treatment for cancer
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-05-19 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Procurement of tissue and blood specimens for research purposes | Up to 5 years
  Tissues and venous blood will be stored, implanted immediately to generate patient-derived xenografts (which require fresh, viable cells), or placed immediately into in vitro cell culture to generate patient-derived cell lines (which require fresh, viable cells).

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, Principal Investigator — National Cancer Institute (NCI)
Locations (140):
- United States (140):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Augusta University Medical Center, Augusta, Georgia
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin